CLINICAL TRIAL: NCT03247218
Title: A Phase - IIa - IIb, Open Label, Single Center Trial to Study the Safety, Tolerability and Efficacy of Memantine Teva® as Supportive Long-term Treatment in Symptomatic Sickle Cell Disease
Brief Title: A Phase - IIa - IIb, Trial to Study the Safety, Tolerability and Efficacy of Memantine as a Long-term Treatment of SCD
Acronym: MeMAGEN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Dr Koren Ariel, Head of Pediatric Hematology Unit, HaEmek Medical Center, Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 071-17 EMC
Record Dates: First submitted 2017-08-01; First posted 2017-08-11 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Memantine

STUDY DESIGN:
Intervention Model Description: a single center and open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single group of patients (Experimental): In this study 40 patients with SCD will be included. Twenty patients aged 18 years or older (cohort 1) and twenty patients 10 - 17 years old (cohort 2).
  All the patients will receive Memantine Teva® film-coated tablets (Memantine hydrochloride) produced by Teva Pharma AG and will be provided as 5 mg, 10 mg, and 20 mg tablets packed in blister.
  The study drug will be taken once a day per os, during one year.
  Interventions: Drug: Memantine Hydrochloride

INTERVENTIONS:
Drug: Memantine Hydrochloride — a low-moderate affinity, uncompetitive, NMDAR antagonist
  Other Names: Memantine TEVA

SUMMARY:
Symptomatic sickle cell disease (SCD) is worldwide the most frequent cause for hereditary hemolytic anemia with recurrent pain crises. Hemolysis, vaso- occlusive and pain crises are hallmarks of this disease and are causative for an important socio-economic burden worldwide, especially in Africa.

Aside from allogenic stem cell transplantation, which is rarely available and very expensive, at present there is no curative treatment for patients with SCD. The current standard of care includes treatment with Hydroxyurea and symptomatic care such as transfusions, antibiotic/analgesic treatment. Recent findings allowed the investigators to come up with a novel pharmacological target for prophylactic treatment of this group of patients. The investigators showed that N-methyl D-aspartate receptors (NMDARs) are substantially up-regulated in circulating red blood cells (RBCs) of SCD patients. Ca2+ uptake via these non-selective cation channels has major impact on RBC hydration and facilitates polymerization of deoxygenated hemoglobin S variant in RBCs of patients. In vitro observations shows that inhibition of NMDARs with Memantine caused re-hydration and largely prevented hypoxia-induced sickling in RBCs. A pilot trial MemSID (NCT02615847) was conducted in August 2015-March 2017 at the Hematology Division of University Hospital Zurich. A small cohort of adult SCD patients was treated with 20 mg Memantine daily to test safety, tolerability and efficacy of this drug and to assess the effect of Memantine on hemolytic activity and RBC stability. Pilot data reveal safety and an impressive therapeutic potential of Memantine in treating SCD patients. Due to a small number of SCD patients in Switzerland, an extended trial including larger number of adult and adolescent patients will be performed at the Pediatric Hematology Unit of the Emek Medical Center in Afula, Israel

DETAILED DESCRIPTION:
Background and Rationale: Symptomatic sickle cell disease (SCD) is worldwide the most frequent cause for hereditary hemolytic anemia with recurrent pain crises. Hemolysis, vaso- occlusive and pain crises are hallmarks of this disease and are causative for an important socio-economic burden worldwide, especially in Africa.

Aside from allogenic stem cell transplantation, which is rarely available and very expensive, at present there is no curative treatment for patients with SCD. The current standard of care includes treatment with Hydroxyurea and symptomatic care such as transfusions, antibiotic/analgesic treatment. Recent findings allowed the investigators to come up with a novel pharmacological target for prophylactic treatment of this group of patients. N-methyl D-aspartate receptors (NMDARs) are substantially up-regulated in circulating red blood cells (RBCs) of SCD patients. Ca2+ uptake via these non-selective cation channels has major impact on RBC hydration and facilitates polymerization of deoxygenated hemoglobin S variant in RBCs of patients. In vitro inhibition of NMDARs with Memantine caused re-hydration and largely prevented hypoxia-induced sickling in RBCs. A pilot trial MemSID (NCT02615847) was conducted in August 2015-March 2017 at the Hematology Division of University Hospital Zurich. A small cohort of adult SCD patients was treated with 20 mg Memantine daily to test safety, tolerability and efficacy of this drug and to assess the effect of Memantine on hemolytic activity and RBC stability. Pilot data reveal safety and an impressive therapeutic potential of Memantine in treating SCD patients. Due to a small number of SCD patients in Switzerland, an extended trial including larger number of adult and adolescent patients will be performed at the Pediatric Hematology Unit of the Emek Medical Center in Afula, Israel.

Objective(s): Primary objective:

To evaluate the safety, tolerability and efficacy of low doses of Memantine Teva® treatment in adult and adolescent patients with symptomatic SCD.

Secondary objective:

To asses and evaluate the long-term effects of Memantine Teva® on the clinical and laboratory parameters in adult and adolescent patients with symptomatic SCD.

The following laboratory parameters will be assessed and evaluated:

* Complete blood count.
* Hemolytic activity (reticulocytes, indirect bilirubin and LDH).
* Iron status (ferritin, serum iron, transferrin and transferrin saturation).
* Fetal hemoglobin levels Additional parameters related to red cell volume, density, membrane stability, adherablilty, inflammatory markers and metabolic activity will be detected by the external laboratory (Red Cell Research Group, University of Zurich) Study design: It is a single center and open label study.

Laboratory analysis including hematology, coagulation and chemistry test will be performed and urine samples will be also analyzed. In addition, at each visit a physical examination and measurement of vital signs will be performed.

The number of total admissions, hospital days and emergency consultations will be recorded. The amount and type of analgesic medication given. The amount of RBC transfusions, the number of days that antibiotics were prescribed will be also recorded.

At screening and at the end of the study SCD specific assessments will be performed, which include cardiologic examination (ECG, ECHO), abdominal sonography, ophthalmological examination, lung function testing and neuroangiologic examination.

The impact on working ability assessed by the number of days with inability to work. For the impact on work ability and social life activities a questionnaire of quality of life will be filled out by the patient once a month.

- Evaluation of Cognitive function will be also performed at screening and at the end of the study Study Product / Intervention: Memantine Teva® is a low-moderate affinity, uncompetitive, NMDAR antagonist and is licensed in Switzerland and in Israel for the treatment of Alzheimer disease.

Memantine Teva® film-coated tablets (Memantine hydrochloride) is produced by Teva Pharma AG and will be provided as 5 mg, 10 mg, and 20 mg tablets packed in blister.

The study drug will be taken once a day per os, during Number of Participants with Rationale: In this study 40 patients with SCD will be included. Twenty patients aged 18 years or older (cohort 1) and twenty patients 10 - 17 years old (cohort 2).

Study Duration: The study lasts 15 month per patient.

ELIGIBILITY:
Inclusion Criteria:

* Documented symptomatic sickle cell disease (HbSS or HbS/beta thalassemia)
* Age 18 years or older (cohort 1) and 10 - 17 years old (cohort 2)
* Able and willing to provide written informed consent and to comply with the study protocol procedures Willing to use two effective methods of contraception during study treatment until 6 months after stop of study treatment. Effective contraception methods are considered oral, injectable, implantative contraceptives or intrauterine contraceptive devices combined with use of condom.

Exclusion Criteria:

* History of transfusion during last three months before Screening
* Patients with active bacterial, viral or fungal infection requiring systemic treatment
* Patients with known infection with human immunodeficiency virus (HIV) of human T cell leukemia virus 1 (HTLV-1)
* Inadequate renal function: creatinine clearance < 30ml/min
* Inadequate liver function: NCICTC Grade 3 liver function tests (AST, ALT > 5x upper limit of normal (ULN))
* Patients with Chronic Active Hepatitis - HCV or HBV
* History of malignancy
* Women who are pregnant or breast feeding
* Known epileptic disease and under treatment with anticonvulsive drugs
* The receipt of any investigational product within 30 days prior to this trial

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-02-02 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of Incidence and severity of Memantine treatment-related Adverse Events (AE), including clinically significant abnormal laboratory values in adult and adolescent patients with symptomatic SCD. | one year
  The following laboratory parameters will be assessed and evaluated:
  * Complete blood count.
  * Hemolytic activity (reticulocytes, indirect bilirubin and LDH).
  * Iron status (ferritin, serum iron, transferrin and transferrin saturation).
  * Fetal hemoglobin levels
  * Red cell volume, density, membrane stability, adherablilty, inflammatory markers and metabolic activity.

SECONDARY OUTCOMES:
Assessment of Clinical Improvement during Memantine treatment compared to a pre-screening data obtained from patients clinical files in adult and adolescent patients with symptomatic SCD. | one year
  Clinical improvements will be assessed by
  * Number of hospital days.
  * Number of emergency consultations
  * Impact on working ability (the number of days with inability to work)
  * The amount and type of analgesic medication received by the patient.
  * The amount of RBC transfusions received by the patient.
  * The number of days that antibiotics were prescribed.
  * A questionnaire on quality of life.
  * Evaluation of Cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Koren, Professor, Principal Investigator — Emek Medical Center
Locations (1):
- Emek Medical Centre, Afula, Israel

IPD SHARING:
Plan to Share IPD: No